CLINICAL TRIAL: NCT04705805
Title: Validation of Two Self-questinnaires on Olfactory Disorders for French Speaking Patients: the Self-evaluation of Olfactory Capacities and Quality of Life Questionnaires
Brief Title: Self-assessment of Olfactory Disorders for French Speaking Patients
Acronym: VIF-DOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7917
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Post-viral Anosmia; Post-traumatic Anosmia; Chronic Rhinosinusitis; Idiopathic Anosmia; Age-related Loss of Smell
Keywords: Olfactory disorders; Self-assessment; Quality of life; Olfactory capacities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patient presenting an olfactory dysfunction of any acquired aetiology that has been evolving for at least 3 months without total recovery.
  Interventions: Behavioral: Self-assessment of olfactory disorders through two questionnaires.
- Control: Patient with no sense of smell problems followed up in ENT for another pathology that does not affect the sense of smell
  Interventions: Behavioral: Self-assessment of olfactory disorders through two questionnaires.

INTERVENTIONS:
Behavioral: Self-assessment of olfactory disorders through two questionnaires. — * Assessment of sense of smell or loss of smell using an Analogue Visual Scale
  * Carrying out the objective smell test (Sniffin' sticks test) (gold standard)
  * Information from two self-questionnaires translated into French: a quality of life questionnaire (The Questionnaire Olfactory Disorders (QOD)) and a self-assessment questionnaire of his olfactory capacities (Self-Mini Olfactory Questionnaire (Self-MOQ))

SUMMARY:
Sense of smell disorders are common and are said to affect up to 20% of the general population. They are often disabling and have a real impact on the quality of life. Smell disorders are most often assessed using a visual analogue scale and more rarely with objective tests (Sniffing Stick Test). Many ENT units do not have these objective tests because they are time-consuming and are not covered by health insurance.

Some teams, such as that of Dr Thomas Hummel of the Carl Gustav Carus University Clinic in Dresden Germany, have developed self-assessment questionnaires for the sense of smell in order to improve the overall care of patients with olfactory disorders. Two of these self-questionnaires seem to us to be particularly relevant for use in everyday practice.

Since then, these questionnaires have already been validated in different languages (English, Chinese, Korean...), but have never been translated and validated in French. Translating and validating these questionnaires into French would make it possible to improve the management and follow-up of French patients with olfactory disorders and to assess the impact of loss of smell on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient affiliated to a sickness insurance social protection scheme, beneficiary or rightful claimant
* Patient who has not expressed his or her opposition to the collection and processing of his or her data for research purposes after the investigator has provided informed information.
* Patient presenting an olfactory dysfunction of any acquired aetiology that has been evolving for at least 3 months without total recovery (case group).
* Patient with no sense of smell problems followed up in ENT for another pathology that does not affect the sense of smell (control group).

Exclusion Criteria:

* Patient in an emergency or life-threatening situation
* Patient under judicial protection
* Patient under guardianship or trusteeship
* Inability to provide informed information to the patient (patient does not speak or understand French)
* Patient with congenital syndromic or non-syndromic congenital anosmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case patients with acquired olfactory disorders will be selected from the ENT primary care clinic of Strasbourg University Hospital.
  Control patient without olfactory disorders are treated for another ENT pathology in the ENT primary care clinic of Strasbourg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Reliability of the self-assessment questionnaire | 3 months
  To assess the reliability of the self-assessment questionnaire of his olfactory capacities (Self-MOQ) in French in patients presenting an olfactory dysfunction of any acquired etiology for more than 3 months using a test-retest trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided